CLINICAL TRIAL: NCT00983008
Title: A Prospective Cohort Study on the Effect and Utilization of Protected Time Among Interns on Extended Duty-Hour Call Shifts
Brief Title: Effect and Utilization of Protected Time Among Interns on Extended Duty-Hour Call Shifts
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too few interns willing to consent to wear the actigraph watches.
Sponsor: Providence Health & Services (Other)
Responsible Party: Principal Investigator, Michelle Schoepflin Sanders, Principal Investigator, Providence Health & Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-085B
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Fatigue; Sleep Deprivation; Depression
Keywords: Signs and Symptoms; Internship and Residency; Fatigue; Medical Errors; Burnout, Professional; Actigraphy; Personnel Staffing and Scheduling; Workload; Adult; Intensive Care Units; Prospective Studies; Work Schedule Tolerance; Disorders of Excessive Somnolence; Guideline Adherence; Internal Medicine Education
MeSH Terms: conditions — Fatigue; Sleep Deprivation; Depression; Signs and Symptoms; Burnout, Professional; Disorders of Excessive Somnolence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Protected Time Group (Experimental): Interns working 30 hour shifts every 3rd night and an average of 80 hours per week in a medical intensive care unit.
  Interventions: Behavioral: Protected time and Dedicated time

INTERVENTIONS:
Behavioral: Protected time and Dedicated time — On Sunday through Thursday nights medical intensive care unit interns will have a 5 hour protected period from 2 to 7 am. During this time they will relinquish their pager and cell phone to the Night Float PGY2 or PGY3 who is already responsible for the ICU patients. The four hours between 2 and 6 am are entirely protected. 6 AM to 7 AM is dedicated time during which the interns will be expected to start pre-rounding on the ICU patients and to begin progress notes for the remaining members of the ICU team but still have no pager, cell phone, or cross coverage duties. On Friday and Saturday nights there will be no protected time but these interns will have 42 consecutive hours off following their extended shifts.
  Other Names: Nap

SUMMARY:
This study will test the feasibility and effectiveness of protected time for physicians in training during 30 hour shifts in a medical intensive care unit. The primary outcome will be fatigue. Secondary outcomes include the amount slept while on call, depression, and burnout.

DETAILED DESCRIPTION:
Background: The Institute of Medicine has proposed 5 hour naps for residents on extended overnight call-duty shifts citing resident and patient safety. Concerns raised about this recommendation include increased handoffs, truncated continuity, and if residents would be able to effectively use the protected time for sleep.

Objectives: The purpose of this study is to test if protected time for sleep during extended duty overnight shifts improves resident fatigue and if they actually utilize the time for sleep.

Methods: All interns rotating through the medical intensive care unit from October 2009 through October 2010 will work extended shifts every 3rd night. On Sunday through Thursday nights they will have a 5 hour protected period from 2 AM to 7 AM. During this time they will relinquish their pager and cell phone to the Night Float PGY2 or PGY3 who is already responsible for the ICU patients. The four hours between 2 and 6 am are entirely protected. From 6 AM to 7 AM, interns will be expected to start computer rounding on the ICU patients and to begin progress notes for the remaining members of the ICU team but still have no pager, cell phone, or cross coverage duties. On Friday and Saturday nights there will be no protected time but these interns will have 42 consecutive hours off following their extended shift.

Results from the October 2009 to October 2010 protected time cohort of interns will be compared with two comparison groups from the same institution and the same medical intensive care unit during the academic year June 2008 to June 2009. The first comparison group is interns working 30 hour shifts every 3rd night without any protected time and an average of 80 hours per week. The second comparison group is interns working a maximum shift length of 16 hours and an average of 60 hours per week.

The primary outcome will be measurement of fatigue (daytime multiple sleep latency tests). Secondary outcomes include the amount slept as measured by actigraphy, assessment of burnout (Maslach Burnout Inventory) and depression (Beck Depression Inventory-II).

ELIGIBILITY:
Inclusion Criteria:

* Interns in the Providence St. Vincent Medical Center Internal Medicine Residency Program who are rotating through the medical intensive care unit.

Exclusion Criteria:

* Refusal to consent to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Fatigue as measured by daytime multiple sleep latency test. | Once, during last week of intervention.

SECONDARY OUTCOMES:
Hours slept during protected time | Once, during last week of intervention
Depression | Once, during last week of intervention
Burnout | Once, during last week of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Dunlap, M.D., Principal Investigator — Internal Medicine Resident Program, Providence St. Vincent Medical Center; Michelle Sanders, M.D., Study Director — Internal Medicine Resident Program, Providence St. Vincent Medical Center; Jay B Ham, M.D., Principal Investigator — Internal Medicine Resident Program, Providence St. Vincent Medical Center; Jeffrely Bluhm, M.D., Study Director — Oregon Pulmonology Associates, Portland, Oregon
Locations (1):
- Providence St. Vincent Medical Center, Portland, Oregon, United States

REFERENCES:
- [Background] Iglehart JK. Revisiting duty-hour limits--IOM recommendations for patient safety and resident education. N Engl J Med. 2008 Dec 18;359(25):2633-5. doi: 10.1056/NEJMp0808736. Epub 2008 Dec 3. No abstract available. PMID 19052119
- [Background] Landrigan CP, Rothschild JM, Cronin JW, Kaushal R, Burdick E, Katz JT, Lilly CM, Stone PH, Lockley SW, Bates DW, Czeisler CA. Effect of reducing interns' work hours on serious medical errors in intensive care units. N Engl J Med. 2004 Oct 28;351(18):1838-48. doi: 10.1056/NEJMoa041406. PMID 15509817
- [Background] Parthasarathy S, Hettiger K, Budhiraja R, Sullivan B. Sleep and well-being of ICU housestaff. Chest. 2007 Jun;131(6):1685-93. doi: 10.1378/chest.06-1398. Epub 2007 Mar 30. PMID 17400688
- [Background] Barger LK, Cade BE, Ayas NT, Cronin JW, Rosner B, Speizer FE, Czeisler CA; Harvard Work Hours, Health, and Safety Group. Extended work shifts and the risk of motor vehicle crashes among interns. N Engl J Med. 2005 Jan 13;352(2):125-34. doi: 10.1056/NEJMoa041401. PMID 15647575
- [Background] Fisman DN, Harris AD, Rubin M, Sorock GS, Mittleman MA. Fatigue increases the risk of injury from sharp devices in medical trainees: results from a case-crossover study. Infect Control Hosp Epidemiol. 2007 Jan;28(1):10-7. doi: 10.1086/510569. Epub 2006 Dec 28. PMID 17230382
- [Background] Fahrenkopf AM, Sectish TC, Barger LK, Sharek PJ, Lewin D, Chiang VW, Edwards S, Wiedermann BL, Landrigan CP. Rates of medication errors among depressed and burnt out residents: prospective cohort study. BMJ. 2008 Mar 1;336(7642):488-91. doi: 10.1136/bmj.39469.763218.BE. Epub 2008 Feb 7. PMID 18258931
- [Background] Lockley SW, Barger LK, Ayas NT, Rothschild JM, Czeisler CA, Landrigan CP; Harvard Work Hours, Health and Safety Group. Effects of health care provider work hours and sleep deprivation on safety and performance. Jt Comm J Qual Patient Saf. 2007 Nov;33(11 Suppl):7-18. doi: 10.1016/s1553-7250(07)33109-7. PMID 18173162
- [Background] Resident duty hours: enhancing sleep, supervision, and safety: Committee on Optimizing Graduate Medical Trainee (Resident) Hours and Work Schedules to Improve Patient Safety. Washington, DC: National Academies Press, 2008. Available online at http://www.nationalacademies.org/morenews/20081202.html . See also Attachment A for a comparison of the ACGME work hours requirements and the recommendations from the Institute of Medicine.
- [Background] Littner MR, Kushida C, Wise M, Davila DG, Morgenthaler T, Lee-Chiong T, Hirshkowitz M, Daniel LL, Bailey D, Berry RB, Kapen S, Kramer M; Standards of Practice Committee of the American Academy of Sleep Medicine. Practice parameters for clinical use of the multiple sleep latency test and the maintenance of wakefulness test. Sleep. 2005 Jan;28(1):113-21. doi: 10.1093/sleep/28.1.113. PMID 15700727
- [Background] Pizza F, Contardi S, Ferlisi M, Mondini S, Cirignotta F. Daytime driving simulation performance and sleepiness in obstructive sleep apnoea patients. Accid Anal Prev. 2008 Mar;40(2):602-9. doi: 10.1016/j.aap.2007.08.014. Epub 2007 Sep 19. PMID 18329412
- [Background] Reddy R, Guntupalli K, Alapat P, Surani S, Casturi L, Subramanian S. Sleepiness in medical ICU residents. Chest. 2009 Jan;135(1):81-85. doi: 10.1378/chest.08-0821. Epub 2008 Nov 18. PMID 19017897
- [Background] Volpp KG, Rosen AK, Rosenbaum PR, Romano PS, Even-Shoshan O, Canamucio A, Bellini L, Behringer T, Silber JH. Mortality among patients in VA hospitals in the first 2 years following ACGME resident duty hour reform. JAMA. 2007 Sep 5;298(9):984-92. doi: 10.1001/jama.298.9.984. PMID 17785643
- [Background] Volpp KG, Rosen AK, Rosenbaum PR, Romano PS, Even-Shoshan O, Wang Y, Bellini L, Behringer T, Silber JH. Mortality among hospitalized Medicare beneficiaries in the first 2 years following ACGME resident duty hour reform. JAMA. 2007 Sep 5;298(9):975-83. doi: 10.1001/jama.298.9.975. PMID 17785642
- [Background] Shetty KD, Bhattacharya J. Changes in hospital mortality associated with residency work-hour regulations. Ann Intern Med. 2007 Jul 17;147(2):73-80. doi: 10.7326/0003-4819-147-2-200707170-00161. Epub 2007 Jun 4. PMID 17548403